CLINICAL TRIAL: NCT03369444
Title: A Phase I/II, Open Label, Multicentre, Ascending Single Dose, Safety Study of a Novel Adeno- Associated Viral Vector (FLT180a) in Patients With Haemophilia B
Brief Title: A Factor IX Gene Therapy Study (FIX-GT)
Acronym: FIX-GT
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Terminated early due to challenges during the COVID-19 pandemic and a change in requirements of data to be submitted for marketing authorisation.
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UCL/15/0552
Record Dates: First submitted 2017-09-13; First posted 2017-12-12 (Actual); Results first posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Hemophilia B
MeSH Terms: conditions — Hemophilia B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- FLT180a, 6x10e^11 vg/kg solution for infusion (Experimental): Participants receiving gene therapy vector at a dose of 6x10e^11 vg/kg
  Interventions: Biological: FLT180a
- FLT180a, 2 x 10e^12 vg/kg solution for infusion (Experimental): Participants receiving gene therapy vector at a dose of 2 x 10e^12 vg/kg
  Interventions: Biological: FLT180a
- FLT180a, 1x10e^12 vg/kg solution for infusion (Experimental): Participants receiving gene therapy vector at a dose of 1 x 10e^12 vg/kg
  Interventions: Biological: FLT180a
- FLT180a, 1.3x10e^12 vg/kg solution for infusion (Experimental): Participants receiving gene therapy vector at a dose of 1.3 x 10e^12 vg/kg
  Interventions: Biological: FLT180a

INTERVENTIONS:
Biological: FLT180a — FLT180a is a replication-incompetent adeno- associated viral vector. The vector is composed of a DNA vector genome encapsidated in an adeno-associated virus derived protein capsid. The expression cassette contains DNA encoding Factor IX.

SUMMARY:
Severe haemophilia B (HB) is a bleeding disorder where a protein made by the body to help make blood clot is either partly or completely missing. This protein is called a clotting factor; with severe haemophilia B, levels of clotting factor IX (FIX) (nine) are very low and affected individuals can suffer life threatening bleeding episodes. HB mainly affects boys and men (normally one in every 30,000 males). Current treatment for HB involves intravenous infusions of factor IX as regular treatment (Prophylaxis) or 'on demand'. On demand treatment is highly effective at stopping bleeding but cannot fully reverse long-term damage that follows after a bleed. Regular treatment can prevent bleeding, however can be invasive for patients and also expensive. This research study aims to test the safety and effectiveness of a gene therapy which produces Factor IX protein in the body. The gene will be given using an inactivated virus called "the vector" ( FLT180a), in a single infusion. The vector has been developed from a virus known as an adeno- associated virus, that has been changed so that it is unable to cause a viral infection in humans. This "inactivated" virus is further altered to carry the Factor IX gene and to make its way within liver cells where Factor IX protein is normally made.

Up to three different doses cohorts of FLT180a will be tested, in up to 24 patients with severe haemophilia B. Patients will be recruited from haemophilia centres in the EU and US. Patients will be in the trial for approximately 40 weeks and will undergo procedures including physical examinations, bloods tests, ECGs and liver ultrasounds.

DETAILED DESCRIPTION:
This was a Phase I/II, open-label, multicentre, ascending single-dose, safety study of FLT180a in patients with severe (FIX activity <1%) or moderately severe (FIX activity 1% to 2% with severe bleeding phenotype) HB. Up to 24 patients were planned to be enrolled; however, the study was terminated early (on 20 October 2020) after 10 patients had been enrolled because of changes to the clinical development plan and recruitment difficulties due to the COVID-19 pandemic.

Patients who provided consent to participate and had historical data on bleeding and FIX consumption documented from the previous 3 years' medical notes were screened for eligibility in this study. During the screening period, patients completed a diary to prospectively record ongoing bleeding events and FIX consumption. Patients were monitored through a comprehensive schedule of safety assessments at outpatient visits for 26 weeks.

On completion of the study, patients are to be followed for 15 years under a separate long term follow-up protocol.

Patients who provided consent to participate in this study underwent screening assessments up to 52 weeks before study Day 0 (FLT180a infusion). Due to the risk of bleeding in this patient population, a washout from the patient's FIX concentrate regimen was not mandated. The investigator was to demonstrate, from the patient's medical records, a documented FIX activity level of <1% for severe patients or <2% for moderately severe patients. If (at the investigator's discretion) a FIX concentrate washout was undertaken during the screening period, a minimum of 5 days' washout was required.

Treatment-eligible patients reported to the study site on the day before receiving the gene therapy infusion (Day 1). On Day 0, FLT180a was administered as a single dose, slow intravenous (IV) infusion into a peripheral vein. The patient remained in the study centre for ≥12 hours and until the investigator deemed the patient fit to be discharged. The first 2 patients treated at each dose level remained at the study centre for 24 hours after infusion before discharge.

Patients who were on prophylactic therapy with FIX concentrates remained on their usual dosing schedule and were closely monitored for FIX activity levels after screening and administration of FLT180a. If FIX activity levels ≥3% were reached, then prophylaxis was held pending a repeat analysis within a period of 72 hours. If the FIX activity levels were ≥3% at that time, then prophylaxis was stopped with continued/regular assessment of FIX activity levels and occurrence of spontaneous bleeding.

Patients were required to undergo study evaluations at intervals over the 26-week, post-treatment period. These evaluations took place either at the study infusion site or at their normal haemophilia treatment centre. To monitor for shedding of vector genome (vg) sequences, patients were required to provide plasma, saliva, urine, stool, and semen samples until the results of 3 successive samples were clear.

This was a first-in-human study; therefore, an ascending-dose design was implemented to enable dose evaluation in a step-wise manner. Three dose cohorts of vector (low, intermediate, and high) were tested in the dose escalation. Two patients were tested at each dose level with an additional patient added in the event of a dose limiting toxicity (DLT) (2 + 1 design). Dose escalation occurred provided there was no more than 1 DLT at any dose cohort and if the resulting FIX activity failed to reach the target level. A reduction of the dose level within a cohort occurred if the FIX activity exceeded defined levels to reduce the risk of exceeding the normal physiological range. A dose reduction occurred when the 2 + 1 design was applied at that new dose level within the cohort. At the discretion of the Sponsor after advice from the trial management group (TMG) and independent data monitoring committee (DMC), additional patients were to be added to any cohort to ensure adequate characterisation of either safety or the FIX response before dose escalation/reductions. The Sponsor, TMG, and DMC planned to select the terminal dose level based on the patient FIX activity levels with the aim of ensuring most patients reached a FIX activity level within normal limits and in the absence of DLTs; the terminal dose level was planned to be expanded to 14 patients, but never reached. This design minimised the number of patients who would need to be dosed at suboptimal levels while allowing evaluation of safety with the option to expand a group on observation of DLTs. An extended 6-week interval was observed between the first and second patient on study to monitor for any unanticipated, delayed adverse events (AEs). Subsequently, when dose escalation was ongoing, the study mandated a minimum 4-week interval between patients during which time efficacy and safety was reviewed before a decision to dose the next patient.

The main risk in this study was a dose-dependent, asymptomatic increase in the serum alanine aminotransferase (ALT) level associated with a decline in FIX levels, suggesting a loss of transduced hepatocytes. In this study, all patients were given a take-home pack of immunosuppressants (prednisolone only) to be taken under the direction of the investigator, which allowed rapid intervention if transaminase elevations were observed. In addition, during the anticipated critical time period all patients were to receive a course of immunosuppressants (prednisolone, methylprednisolone, and tacrolimus) beginning at the Week 3 visit or Week 4 visit in line with the relevant protocol version active at the time.

The main efficacy endpoint was based on an analysis of the proportion of patients achieving a clinical or normalised FIX response at 26 weeks. A clinical FIX response was defined as achieving a FIX activity of 5% to 150% of normal. Five percent had been selected as the threshold for a clinical FIX response because using gene therapy in patients with HB to increase FIX activity from <1% to 5% had previously been shown to lead to a highly clinically significant improvement in annualised bleeding rates (ABR) and exogenous factor consumption. A normalised FIX response was defined as achieving a FIX activity level in the normal range (50% to 150%). The normal range had been selected as the threshold level for a normalised FIX response because reaching this level was expected to modify the patient phenotype from severe at study start to normal at which point patients would not be expected to experience spontaneous bleeds.

The choice of a 26-week endpoint was based on previous experience with Adeno-Associated Virus (AAV) gene therapy for HB in which patients achieved steady-state FIX levels by 16 weeks after gene therapy. Based on this, it was anticipated that the patients' FIX activity would reach a stable level by 26 weeks, thus this was an appropriate point at which to measure activity.

ELIGIBILITY:
Inclusion Criteria:

1. Adults males, ≥ 18 years of age.
2. Confirmed diagnosis of HB defined as one of the following:

   1. Documented severe FIX deficiency with plasma FIX activity of <1% of normal, or
   2. moderately severe FIX deficiency with plasma FIX activity level between ≥1% and ≤2% and a severe bleeding phenotype defined by one of the following: i. On prophylaxis for a history of bleeding, or ii. On demand therapy with a history of 4 or more bleeding episodes/year on average over the past 3 years, or iii. evidence of chronic haemophilic arthropathy (pain, joint destruction, and loss of range of motion).
3. Able to give full informed consent and able to comply with all requirements of the trial including 15-year long-term follow-up.
4. Willing to practice barrier contraception until at least 3 consecutive semen samples after vector administration are negative for vector sequences.
5. Lack of neutralising anti-AAV-S3 antibodies using an in vivo transduction inhibition assay within 4 weeks of vector administration.
6. At least 150 exposure days to FIX concentrates.

Exclusion Criteria:

1. Presence of neutralising anti-human FIX antibodies (inhibitor, determined by the Bethesda inhibitor assay) at the time of enrolment or a previous history of FIX inhibitor;
2. Patients at high risk of thromboembolic events (high risk patients would include those with a history of arterial or venous thromboembolism (e.g. deep vein thrombosis, pulmonary embolism, non-haemorrhagic stroke, arterial embolus) and those with acquired thrombophilia including conditions such as atrial fibrilation);
3. Use of investigational therapy for haemophilia within 30 days before enrolment;
4. Patients with active hepatitis B or C, and hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) Ribonucleic acid (RNA) viral load positivity, respectively, or currently on antiviral therapy for hepatitis B or C. Negative viral assays in 2 samples, collected at least 6 months apart, will be required to be considered negative. Both natural clearers and those who have cleared HCV on antiviral therapy are eligible.;
5. Serological evidence of human immunodeficiency virus (HIV-1);
6. Evidence of liver dysfunction (persistently elevated alanine aminotransaminase, aspartate aminotransferase, bilirubin >1.5 x upper limit of normal);
7. Platelet count <50 x 109/L;
8. Uncontrolled glaucoma, diabetes mellitus, or hypertension;
9. Malignancy requiring treatment;
10. Patients with uncontrolled cardiac failure, unstable angina or myocardial infarction in the past 6 months;
11. Poor performance status (World Health Organization score >1);
12. Prior treatment with any gene transfer medicinal product;
13. Known or suspected intolerance, hypersensitivity or contraindication to the investigational product and non-investigational medicinal products or their excipients;
14. Planned major elective surgery prior to the end of trial.
15. Current or relevant history of a physical or psychiatric illness or any medical condition that in the opinion of the investigator could affect the patients safety or interfere with the study assessments.
16. Cytomegalovirus (CMV) Immunoglobulin G (IgG) positive patients who are CMV PCR positive at screening.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pratima Chowdary, Principal Investigator — University College London / Royal Free London NHS Foundation Trust
Locations (11):
- St Jude Children's Research Hospital, Memphis, Tennessee, United States
- St James's Hospital, Dublin, Ireland
- University of Milan, Milan, Italy
- United Kingdom (8):
  - Basingstoke Haemostasis and Thrombosis Centre, Basingstoke
  - East Kent Hospitals University, Canterbury
  - Guy's and St Thomas's NHS Foundation Trust, London
  - Royal Free Hospital, London
  - Newcastle Hospitals NHS Trust, Newcastle upon Tyne
  - Oxford University Hospital, Oxford
  - University of Sheffield, Sheffield
  - University Hospital Southampton, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chowdary P, Shapiro S, Makris M, Evans G, Boyce S, Talks K, Dolan G, Reiss U, Phillips M, Riddell A, Peralta MR, Quaye M, Patch DW, Tuddenham E, Dane A, Watissee M, Long A, Nathwani A. Phase 1-2 Trial of AAVS3 Gene Therapy in Patients with Hemophilia B. N Engl J Med. 2022 Jul 21;387(3):237-247. doi: 10.1056/NEJMoa2119913. PMID 35857660

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All patients enrolled were dosed. There are no significant events in the study that occur between enrolment and dosing.
Groups:
- FLT180a First Dose: 6x10e^11 vg/kg solution for infusion
- FLT180a Second Dose: 2x10e^12 vg/kg solution for infusion
- FLT180a Third Dose: 1x10e^12 vg/kg solution for infusion
- FLT180a Fourth Dose: 1.3x10e^12 vg/kg solution for infusion
Period: Overall Study
Arm/Group | FLT180a First Dose | FLT180a Second Dose | FLT180a Third Dose | FLT180a Fourth Dose
Started | 2 | 2 | 2 | 4
Completed | 2 | 2 | 2 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- FLT180a Fourth Dose: 1.3x10e11 vg/kg solution for infusion
- Total: Total of all reporting groups
Arm/Group | FLT180a First Dose | FLT180a Second Dose | FLT180a Third Dose | FLT180a Fourth Dose | Total
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 10
Age, Customized [Count of Participants; unit: Participants]
  Between 18 and 67 years | 2 | 2 | 2 | 4 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 2 | 2 | 2 | 4 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 2 | 4 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 2 | 2 | 2 | 3 | 9
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 2 | 2 | 2 | 4 | 10
Body Mass Index [Mean (Full Range); unit: kg/m2] | 21.3 [21.2 to 21.4] | 29.55 [27.0 to 32.1] | 24.75 [23.0 to 26.5] | 28.75 [25.2 to 31.0] | 26.62 [21.2 to 32.1]

OUTCOME MEASURES:

1. Primary Outcome: Frequency and Severity of Treatment-emergent Adverse Events (TEAEs) (Safety)
Description: Safety as assessed by the reporting of AEs according to Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Time Frame: From Day 0 (first dose of FLT180a) until week 26 post infusion (up to 26 weeks)
Population: All treated patients.
Measure: Number; unit: Events
Arm/Group | FLT180a First Dose | FLT180a Second Dose | FLT180a Third Dose | FLT180a Fourth Dose
Number analyzed (Participants) | 2 | 2 | 2 | 4
Events
  Number of TEAEs | 11 | 37 | 25 | 108
  Serious TEAEs | 0 | 6 | 4 | 5
  FLT180a-related TEAEs | 0 | 13 | 4 | 10
  Serious FLT180a-related TEAEs | 0 | 3 | 4 | 4

2. Primary Outcome: Number of Participants With FIX Activity Response
Description: The proportion of participants at the terminal dose (1.3 x 10e^12 vg/kg) achieving clinical FIX response and proportion of patients achieving normalised FIX response at Week 26. A clinical FIX response is defined as achieving a FIX activity of 5% to 150%. Normalised FIX response is defined as achieving FIX activity in the normal range (50-150%).
Time Frame: From screening until week 26 post infusion (Up to 38 weeks)
Population: Patients treated at the terminal dose (1.3x10e12 vg/kg)
Measure: Count of Participants; unit: Participants
Arm/Group | FLT180a Fourth Dose
Number analyzed (Participants) | 4
Participants
  Clinical FIX Responders (≥5% and ≤150% of Normal) | 2
  Normalised FIX Responders (≥50% and ≤150% of Normal) | 2

3. Secondary Outcome: Number of Participants With a Change From Baseline or Abnormal Finding From Routine Safety Assessments
Description: Safety as assessed by reporting of abnormal or change from baseline findings from routine safety assessments including, laboratory assessments, ECG, physical exam and liver ultrasound.
Time Frame: From screening until week 26 post infusion (Up to 38 weeks)
Population: Safety as assessed by reporting of abnormal or change from baseline findings from safety assessments including, laboratory assessments, vital signs, ECG, physical exam and liver ultrasound.
Measure: Number; unit: Number of participants
Arm/Group | FLT180a First Dose | FLT180a Second Dose | FLT180a Third Dose | FLT180a Fourth Dose
Number analyzed (Participants) | 2 | 2 | 2 | 4
Number of participants
  Haemoglobin | 0 | 1 | 0 | 2
  Leukocytes (10e9/L0 | 1 | 0 | 2 | 1
  Lymphocytes count decreased (10e9/L) | 1 | 2 | 2 | 3
  Lymphocytes count increased (10e9/L) | 0 | 0 | 0 | 2
  Neutrophils (10e9/L) | 1 | 0 | 0 | 1
  Platelets (10e9/L) | 1 | 1 | 1 | 0
  Basophils (10e9/L) | 0 | 0 | 0 | 0
  Eosinophils (10e9/L) | 0 | 0 | 0 | 0
  Erythrocytes (10e12/L) | 1 | 2 | 2 | 2
  Hemotocrit (L/L) | 0 | 1 | 0 | 1
  Monocytes (10e9/L) | 1 | 2 | 0 | 1
  Thrombin/Antithrombin (ug/L) | 2 | 2 | 2 | 4
  Alanine Aminotransferase (U/L) | 0 | 1 | 1 | 2
  Albumin (g/L) | 0 | 0 | 0 | 0
  Alkaline Phosphatase (U/L) | 0 | 0 | 0 | 0
  Aspartate Aminotransferase (U/L) | 0 | 1 | 0 | 3
  Bilirubin (umol/L) | 1 | 0 | 0 | 0
  Creatinine (umol/L) | 2 | 1 | 1 | 2
  Glucose (mmol/L) | 1 | 2 | 0 | 0
  Potassium (mmol/L) (Hyperkalemia) | 0 | 0 | 0 | 1
  Potassium (mmol/L) (Hypokalemia) | 0 | 1 | 0 | 0
  Sodium (mml/L) (Hypernatremia) | 0 | 0 | 0 | 1
  Sodium (mml/L) (Hyponatremia) | 0 | 1 | 0 | 1
  BiCarbonate (mmol/L) | 1 | 2 | 2 | 4
  C Reactive Protein (mg/L) | 0 | 1 | 1 | 4
  Chloride (mmol/L) | 2 | 2 | 0 | 1
  Direct Bilirubin (umol/L) | 1 | 0 | 0 | 0
  Indirect Billirubin (umol/L) | 1 | 0 | 0 | 0
  Phosphate (mmol/L) | 2 | 1 | 1 | 4
  Protein (g/L) | 1 | 1 | 1 | 3
  Urea Nitrogen (mmol/L) | 0 | 1 | 1 | 3
  ECG Overall Shift from Baseline | 0 | 1 | 1 | 1
  Physical Exam - Head - Week 16 post dose abnormal - Not clinically Significant (NCS) | 0 | 0 | 1 | 0
  Physical Exam - Head - Week 20 post dose abnormal NCS | 0 | 0 | 1 | 0
  Physical Exam - Neck - Week 14 post dose abnormal -Clinically Significant (CS) | 0 | 0 | 0 | 2
  Physical Exam - Eyes - Week 14 post dose abnormal NCS | 0 | 0 | 0 | 1
  Physical Exam - Ears, Nose, Throat - Week 12 post dose abnormal NCS | 0 | 0 | 0 | 1
  Physical Exam - Chest - Week 2 post dose abnormal NCS | 0 | 0 | 0 | 1
  Physical Exam - Heart - Week 11 post dose abnormal NCS | 0 | 1 | 0 | 0
  Physical Exam - Heart - Week 16 post dose abnormal CS | 0 | 0 | 0 | 1
  Physical Exam - Heart - Week 20 post dose abnormal NCS | 0 | 0 | 0 | 1
  Physical Exam - Abdomen - Week 1 post dose abnormal NCS | 0 | 1 | 0 | 0
  Physical Exam - Abdomen - Week 2 post dose abnormal NCS | 0 | 1 | 0 | 0
  Physical Exam - Abdomen - Week 3 post dose abnormal NCS | 0 | 1 | 0 | 0
  Physical Exam - Abdomen - Week 4 post dose abnormal NCS | 0 | 1 | 0 | 0
  Physical Exam - Abdomen - Week 5 post dose abnormal NCS | 0 | 1 | 0 | 0
  Physical Exam - Abdomen - Week 6 post dose abnormal NCS | 0 | 1 | 0 | 0
  Physical Exam - Abdomen - Week 7 post dose abnormal NCS | 0 | 1 | 0 | 0
  Physical Exam - Abdomen - Week 8 post dose abnormal NCS | 0 | 1 | 0 | 0
  Physical Exam - Abdomen - Week 9 post dose abnormal NCS | 0 | 1 | 0 | 0
  Physical Exam - Abdomen - Week 10 post dose abnormal NCS | 0 | 1 | 0 | 0
  Physical Exam - Abdomen - Week 11 post dose abnormal NCS | 0 | 1 | 0 | 0
  Physical Exam - Skin - Week 2 post dose abnormal NCS | 0 | 0 | 1 | 0
  Physical Exam - Skin - Week 3 post dose abnormal NCS | 0 | 0 | 1 | 0
  Physical Exam - Skin - Week 4 post dose abnormal NCS | 0 | 1 | 0 | 0
  Physical Exam - Skin - Week 5 post dose abnormal NCS | 0 | 1 | 1 | 0
  Physical Exam - Skin - Week 6 post dose abnormal NCS | 0 | 1 | 1 | 0
  Physical Exam - Skin - Week 7 post dose abnormal NCS | 0 | 0 | 2 | 1
  Physical Exam - Skin - Week 8 post dose abnormal NCS | 0 | 1 | 2 | 0
  Physical Exam - Skin - Week 9 post dose abnormal NCS | 0 | 1 | 1 | 1
  Physical Exam - Skin - Week 9 post dose abnormal CS | 1 | 0 | 1 | 0
  Physical Exam - Skin - Week 10 post dose abnormal NCS | 0 | 1 | 2 | 1
  Physical Exam - Skin - Week 11 post dose abnormal NCS | 0 | 0 | 0 | 1
  Physical Exam - Skin - Week 11 post dose abnormal CS | 0 | 0 | 2 | 0
  Physical Exam - Skin - Week 12 post dose abnormal NCS | 0 | 0 | 0 | 1
  Physical Exam - Skin - Week 12 post dose abnormal CS | 0 | 0 | 2 | 0
  Physical Exam - Skin - Week 14 post dose abnormal CS | 0 | 0 | 2 | 0
  Physical Exam - Skin - Week 16 post dose abnormal NCS | 0 | 0 | 0 | 1
  Physical Exam - Skin - Week 20 post dose abnormal NCS | 0 | 0 | 1 | 1
  Physical Exam - Neurological Systems - Week 1 post dose abnormal NCS | 0 | 1 | 0 | 0
  Physical Exam - Neurological Systems - Week 2 post dose abnormal NCS | 0 | 1 | 0 | 0
  Physical Exam - Neurological Systems - Week 3 post dose abnormal NCS | 0 | 1 | 0 | 0
  Physical Exam - Neurological Systems - Week 4 post dose abnormal NCS | 0 | 1 | 0 | 1
  Physical Exam - Neurological Systems - Week 5 post dose abnormal NCS | 0 | 1 | 0 | 0
  Physical Exam - Neurological Systems - Week 5 post dose abnormal CS | 0 | 0 | 0 | 1
  Physical Exam - Neurological Systems - Week 6 post dose abnormal NCS | 0 | 1 | 0 | 0
  Physical Exam - Neurological Systems - Week 6 post dose abnormal CS | 0 | 0 | 0 | 1
  Physical Exam - Neurological Systems - Week 7 post dose abnormal NCS | 0 | 1 | 0 | 0
  Physical Exam - Neurological Systems - Week 7 post dose abnormal CS | 0 | 0 | 0 | 1
  Physical Exam - Neurological Systems - Week 8 post dose abnormal NCS | 0 | 1 | 0 | 0
  Physical Exam - Neurological Systems - Week 8 post dose abnormal CS | 0 | 0 | 0 | 2
  Physical Exam - Neurological Systems - Week 9 post dose abnormal NCS | 0 | 1 | 0 | 0
  Physical Exam - Neurological Systems - Week 9 post dose abnormal CS | 0 | 0 | 0 | 2
  Physical Exam - Neurological Systems - Week 10 post dose abnormal CS | 0 | 0 | 0 | 1
  Physical Exam - Neurological Systems - Week 11 post dose abnormal NCS | 0 | 1 | 0 | 1
  Physical Exam - Neurological Systems - Week 11 post dose abnormal CS | 0 | 0 | 0 | 1
  Physical Exam - Neurological Systems - Week 12 post dose abnormal NCS | 0 | 0 | 0 | 1
  Physical Exam - Neurological Systems - Week 12 post dose abnormal CS | 0 | 0 | 0 | 1
  Physical Exam - Neurological Systems - Week 14 post dose abnormal NCS | 0 | 1 | 0 | 1
  Physical Exam - Neurological Systems - Week 14 post dose abnormal CS | 0 | 0 | 0 | 1
  Physical Exam - Neurological Systems - Week 16 post dose abnormal NCS | 0 | 1 | 0 | 1
  Physical Exam - Neurological Systems - Week 16 post dose abnormal CS | 0 | 0 | 0 | 1
  Physical Exam - Neurological Systems - Week 20 post dose abnormal NCS | 0 | 1 | 0 | 0
  Physical Exam - Neurological Systems - Week 20 post dose abnormal CS | 0 | 0 | 0 | 1
  Physical Exam - Neurological Systems - Week 26/EOS post dose abnormal NCS | 0 | 1 | 0 | 1
  Physical Exam - Lung - Week 7 post dose abnormal CS | 0 | 0 | 0 | 1

4. Secondary Outcome: FIX Concentrate Usage
Description: Change from baseline in FIX concentrate consumption.
Time Frame: Baseline and Post Dose (Day15 post infusion to Week26/End of Study)
Measure: Mean (Standard Deviation); unit: International Units (IU)
Groups:
- FLT180a First Dose: Dose 6x10e^11 vg/kg Solution for infusion
- FLT180a Second Dose: Dose 2x10e^12 vg/kg solution for infusion
Arm/Group | FLT180a First Dose | FLT180a Second Dose | FLT180a Third Dose | FLT180a Fourth Dose
Number analyzed (Participants) | 2 | 2 | 2 | 4
International Units (IU)
  Annualised Total Units (IU) of FIX Concentrate Consumption at Baseline | 501500 (300520.38) | 1219000 (72124.89) | 968000 (14142.14) | 350947.5 (112653.53)
  Annualised Total Total Units (IU) of FIX Concentrate Consumption Post-Dose (Day 15 to Week 26/EOS) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

5. Secondary Outcome: Bleeding Frequency
Description: Change from baseline in annualised bleeding rate (ABR)
Time Frame: Baseline and Post-Dose (Day 15 to Week 26/EOS)
Measure: Mean (Standard Deviation); unit: Bleeds per year
Arm/Group | FLT180a First Dose | FLT180a Second Dose | FLT180a Third Dose | FLT180a Fourth Dose
Number analyzed (Participants) | 2 | 2 | 2 | 4
Bleeds per year
  ABR at Baseline (over last 3 years) | 4.665 (0.9405) | 4.330 (4.2426) | 1.0 (1.4142) | 2.335 (1.1208)
  ABR at Post-Dose (Day 15 to WEek 26/EOS) | 2.175 (3.0759) | 0 (0) | 2.160 (3.0547) | 0.548 (1.0950)

6. Secondary Outcome: Immune Response - Development of Inhibitors
Description: Immune response to the human FIX transgene product (i.e., development of FIX neutralising antibodies referred to as inhibitors) will be assessed by measurement of the level of inhibitors.
Time Frame: Week 1, week 2, week 3, week 6, week 9, week 12, week 16, week 20 and week 26/EOS post infusion
Population: Immune response to the FIX transgene product (ie, development of inhibitors) was assessed by measurement of the level of inhibitors. The FIX inhibitor titre results could not be quantified accurately where a participants basal FIX activity was >20%. Where this occurred the FIX inhibitor values could not be measured and was deemed missing.
Measure: Count of Participants; unit: Participants
Arm/Group | FLT180a First Dose | FLT180a Second Dose | FLT180a Third Dose | FLT180a Fourth Dose
Number analyzed (Participants) | 2 | 2 | 2 | 4
Participants
  Week 1: <0.4 BU | 1 | 0 | 2 | 0
  Week 1: Missing | 1 | 2 | 0 | 4
  Week 2: <0.4 BU | 2 | 0 | 2 | 0
  Week 2: Missing | 0 | 2 | 0 | 4
  Week 3: <0.4 BU | 1 | 0 | 0 | 0
  Week 3: Missing | 1 | 2 | 2 | 4
  Week 6: <0.4 BU | 0 | 0 | 1 | 0
  Week 6: Missing | 2 | 2 | 1 | 4
  Week 9: <0.4 BU | 0 | 0 | 0 | 0
  Week 9: Missing | 2 | 2 | 2 | 4
  Week 12: <0.4 BU | 0 | 0 | 0 | 0
  Week 12: Missing | 2 | 2 | 2 | 4
  Week 16: <0.4 BU | 0 | 0 | 0 | 0
  Week 16: Missing | 2 | 2 | 2 | 4
  Week 20: <0.4 BU | 0 | 0 | 0 | 0
  Week 20: Missing | 2 | 2 | 2 | 4
  Week 26/EOS: <0.4 BU | 0 | 0 | 1 | 0
  Week 26/EOS: Missing | 2 | 2 | 1 | 4

7. Secondary Outcome: Viral Shedding Evaluated as Time to Unquantifiable Vector Genomes
Description: Serum and bodily secretions will be collected to assess clearance of vector genomes
Time Frame: From screening until time to unquantifiable results of vector genomes in all matrices, up to an average of 5.14 weeks
Population: Vector Genomes in Plasma, Saliva, Urine, Stool and Semen: Time to unquantifiable results (weeks)
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | FLT180a First Dose | FLT180a Second Dose | FLT180a Third Dose | FLT180a Fourth Dose
Number analyzed (Participants) | 2 | 2 | 2 | 4
Weeks
  Plasma | 1.355 (1.1102) | 1.715 (0.6010) | 1.425 (1.0112) | 1.750 (0.6320)
  Saliva | 0.570 (0.000) | 2.570 (0.6081) | 1.355 (1.1102) | 2.143 (0.9972)
  Semen | 2.285 (0.2051) | 3.070 (0.0990) | 2.640 (0.7071) | 3.750 (1.0357)
  Stool | 2.930 (0.7071) | 4.290 (1.4142) | 5.140 (1.4142) | 3.788 (0.5007)
  Urine | 1.355 (1.1102) | 2.070 (0.0990) | 2.140 (0.0000) | 1.178 (0.7590)

8. Secondary Outcome: Endogenous FIX Production
Description: The proportion of patients achieving FIX activity at or above 5%, 15%, 30%, 40%, 50%, 70% and 150% of normal, at each scheduled visit, will be summarised by dose and overall.
Time Frame: From screening until week 26 post infusion
Population: Endogenous FIX production at visit week 26/EOS
Measure: Number; unit: Number of participants
Groups:
- FLT180a First Dose: 6x10e11 vg/kg solution for infusion
- FLT180a Second Dose: 2x10e12 vg/kg solution for infusion
- FLT180a Third Dose: 1x10e12 vg/kg solution for infusion
- FLT180a Forth Dose: 1.3x10e12 vg/kg solution for infusion
Arm/Group | FLT180a First Dose | FLT180a Second Dose | FLT180a Third Dose | FLT180a Forth Dose
Number analyzed (Participants) | 2 | 2 | 2 | 4
Number of participants
  FIX Activity ≥5% and ≤150% of Normal | 2 | 1 | 2 | 2
  FIX Activity ≥15% and ≤150% of Normal | 2 | 1 | 1 | 2
  FIX Activity ≥30% and ≤150% of Normal | 2 | 1 | 1 | 2
  FIX Activity ≥40% and ≤150% of Normal | 2 | 1 | 1 | 2
  FIX Activity ≥50% and ≤150% of Normal | 0 | 1 | 1 | 2
  FIX Activity ≥70% and ≤150% of Normal | 0 | 1 | 0 | 1
  FIX Activity ≥5% of Normal | 2 | 2 | 2 | 4
  FIX Activity ≥15% of Normal | 2 | 2 | 1 | 4
  FIX Activity ≥30% of Normal | 2 | 2 | 1 | 4
  FIX Activity ≥40% of Normal | 2 | 2 | 1 | 4
  FIX Activity ≥50% of Normal | 0 | 2 | 1 | 4
  FIX Activity ≥70% of Normal | 0 | 2 | 0 | 3

9. Secondary Outcome: Change From Baseline in FIX Activity as a Percentage of Normal Values
Description: Absolute change from baseline in FIX production (% FIX activity) at week 26/EOS will be summarised.
Time Frame: Week 26/EOS
Population: Absolute change from baseline in FIX production (% FIX activity) at week 26/EOS
Measure: Mean (Standard Deviation); unit: FIX Activity (%)
Arm/Group | FLT180a First Dose | FLT180a Second Dose | FLT180a Third Dose | FLT180a Fourth Dose
Number analyzed (Participants) | 2 | 2 | 2 | 4
FIX Activity (%) | 40 (7.07) | 155.5 (157.68) | 32.0 (41.01) | 129.3 (65.7)

ADVERSE EVENTS:
Time Frame: From consent to Week 26 post dose/End of Study visit or early withdrawal of patient (up to 38 weeks).
Description: Any untoward medical occurrence in a clinical investigation subject administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment.
Groups:
- FLT180a Forth Dose: 1.3x10e^12 vg/kg solution for infusion
Arm/Group | FLT180a First Dose | FLT180a Second Dose | FLT180a Third Dose | FLT180a Forth Dose
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/2 | 2/2 | 2/2 | 3/4
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 2/2 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FLT180a First Dose (N=2) | FLT180a Second Dose (N=2) | FLT180a Third Dose (N=2) | FLT180a Forth Dose (N=4)
Increased ALT (Investigations) | 0 (0) | 2 (2) | 2 (3) | 0 (0) — Alanine aminotransferase increased
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Epigastric Pain
Raised Troponin (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Raised Troponin
Raised Amylase (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Amylase increased
Chest Sepsis (no more information) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Pulmonary sepsis
Drop in Factor IX (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Coagulation factor IX level decreased
Transaminitis (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (4) — Transaminases increased
Tacrolimus Toxicity (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Toxicity to various agents
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FLT180a First Dose (N=2) | FLT180a Second Dose (N=2) | FLT180a Third Dose (N=2) | FLT180a Forth Dose (N=4)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (5) | 2 (3) | 2 (2)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Coagulation factor IX level increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coagulation factor IX level decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug level increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 3 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (2) | 1 (3) | 3 (8)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (2) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (5)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (10)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Burning sensation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Bladder pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cushingoid (Endocrine disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Protocol defined number of participants (n=24) was not met, the terminal dose as specified in the protocol was not identified prior to early study termination.

The primary efficacy endpoints (FIX response at the terminal dose) could therefore not be detailed established. However the FIX response data (efficacy endpoint) for the 4 patients treated at the last studied dose level 1.3×10e^12 vg/kg, have been presented instead.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-04-21): https://cdn.clinicaltrials.gov/large-docs/44/NCT03369444/Prot_001.pdf
  • Statistical Analysis Plan (2021-01-29): https://cdn.clinicaltrials.gov/large-docs/44/NCT03369444/SAP_002.pdf